CLINICAL TRIAL: NCT06863233
Title: Assessment of Patients Immune Response After Treatment With Engineered Tumor Infiltrating Lymphocyte Therapy Incorporating CD8 PET Imaging
Brief Title: A Study of CD8+ T Cell Imaging During Treatment in People With Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-369
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer; Metastatic Non Small Cell Lung Cancer
Keywords: Lung Cancer; Non Small Cell Lung Cancer; Metastatic Non Small Cell Lung Cancer; Memorial Sloan Kettering Cancer Center; 24-369
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Metastatic non-small cell lung cancer (NSCLC) (Experimental): Participants will have a diagnosis of metastatic non-small cell lung cancer (NSCLC)
  Interventions: Drug: Zirconium Zr 89 crefmirlimab berdoxam; Diagnostic Test: PET/CT Scan

INTERVENTIONS:
Drug: Zirconium Zr 89 crefmirlimab berdoxam — Zirconium Zr 89 crefmirlimab berdoxam, the investigational agent proposed in this imaging study, is an anti-CD8 minibody (crefmirlimab), conjugated with deferoxamine (Df, berdoxam) and radiolabeled with Zirconium-89.
Diagnostic Test: PET/CT Scan — Each patient will undergo up to four infusions of Zirconium Zr 89 crefmirlimab berdoxam followed by PET/CT 24 hours later (+/- 3 hours).

SUMMARY:
The purpose of this study to learn whether PET/CT (positron emission tomography/computed tomography) scans using an imaging agent (radiotracer) called zirconium Zr 89 crefmirlimab berdoxam is a safe and effective way to identify CD8+ T cells

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older at the time of signing the informed consent.
* Patient has a histologically confirmed diagnosis of metastatic non-small cell lung cancer
* Patient is enrolled in the engineered TIL cell therapy protocol OBX115-23-01, but has not received the treatment yet.
* Men and women of child-producing potential, use of effective double barrier contraceptive methods during the study, up to 30 days after the last administration of the investigational product.
* Patient or legally authorized representative provided signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Patient or legally authorized representative provided written authorization for use and disclosure of protected health information.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients with a history of splenectomy or significant splenic dysfunction (e.g., as evidenced by splenomegaly or a history of recurrent infections due to impaired immune function)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2028-03-03 (Estimated); Study Completion 2028-03-03 (Estimated)

PRIMARY OUTCOMES:
Difference between Zirconium Zr 89 crefmirlimab berdoxam PET uptake at pre- vs post-TIL infusion and pre- vs post-ACZ redosing. | Baseline to two weeks
  Assess the distribution of the CD8+ cells during TIL therapy by measuring the largest difference in Zirconium Zr 89 crefmirlimab berdoxam PET uptake at pre- vs post-TIL infusion and pre- vs post-ACZ redosing.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Schoenfeld, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activities), New York, New York
  - Memorial Sloan Kettering Cancer Center @ Nassau (Consent only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org